CLINICAL TRIAL: NCT07143565
Title: Chat-based Text Messaging and Online Education Hubs for Reducing Alcohol Consumption and Binge Drinking in Adolescents: A Pilot Randomized Controlled Trial
Brief Title: Online Education Hubs and Chat-based Text Messaging for Reducing Alcohol Consumption and Binge Drinking in Adolescents: A Pilot Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: knowledgehub
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Teen Drinking
Keywords: Gamification; Information Hub; Randomized Controlled Trial; Teen Drinking; Binge Drinking
MeSH Terms: conditions — Underage Drinking; Binge Drinking

STUDY DESIGN:
Intervention Model Description: 2-arm: Intervention group and Control group
Masking Description: open-labelled RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The treatment package includes both optional and mandatory treatments. The mandatory treatments consist of mHealth text messaging and an online platform hub.
  Interventions: Behavioral: Online platform hub and mHealth Text Messaging
- Control Group (Active Comparator): The control group will be provided a self-help material like leaflet for alcohol reduction, which involves education on alcohol harm and strategies for alcohol reduction.
  Interventions: Behavioral: Self-help material

INTERVENTIONS:
Behavioral: Online platform hub and mHealth Text Messaging — The treatment package includes both optional and mandatory treatments. The mandatory treatments consist of mHealth text messaging and an online platform hub. We have developed a game which educates teenagers about alcohol reduction and promotes awareness of alcohol-related harm. Designed to be both engaging and informative, the game uses real-life scenarios, interactive storytelling, and decision-based gameplay to help young people understand the risks of excessive drinking. Also, participants with Audit Score > 7 will receive individualized chat-based instant text messages from WhatsApp for 8 weeks. They will have real-time and one-to-one interaction. The conversation intensity depends on the participants' need.
  Arms: Intervention group
Behavioral: Self-help material — Self-help material like leaflet is a common method used in preventing teenage Drinking.
  Arms: Control Group

SUMMARY:
Online education hubs and Chat-based text messaging for reducing alcohol consumption and binge drinking in adolescents: A pilot randomized controlled trial

DETAILED DESCRIPTION:
It is urged to alleviate the problem before it become worse. Department of Health in Hong Kong developed 3 information hubs (Alcohol Fails, Young and Alcohol Free and Understanding Alcohol Harm) to distribute alcohol-related messages, such as binge drinking. Yet, it lacks interactive and individualized elements, which makes it difficult to attract secondary school students to search for information. Our previous research also reveals that more than 80% of the respondents are willing to receive message reminders for controlling or avoiding binge drinking. They also suggest that those messages should include drinking limits, health risks, psychological support, and alternative activities. It proves that an interactive and personalized intervention package should be included in secondary school in terms of binge drinking prevention. This could be a research gap to investigate in this project.

We expect that this study result would demonstrate the main effects of the interventions, including mHealth text messaging, and online platform hub. By analyzing those intervention results, we could deeply understand the effective methods to lower the risk of young adult binge drinking phenomenon. We could provide more precise interventions to secondary school students. This study will also prepare for future RCTs to explore the possibility on the integration of other intervention components or factors for binge drinking prevention research. In the long run, the proportion of binge drinking in population and young-aged will be lowered. Department of Health or other future research could implement this intervention as a fundamental to enhance the effectiveness of the alcohol control intervention.

A pilot 2-arm, parallel, open-labelled randomized controlled trial randomly allocated participants (1:1 ratio) to intervention and control groups. The intervention group has 2 intervention components: (1) Online information hub (compulsory: game), (2) mHealth text messaging at last to people who needed (Audit score >7). The control group will receive self-help materials during the same period. The sample size is 100 participants (50 for each group).

100 ever-drinkers will be recruited from the secondary schools through online and offline. Study information will be disseminated via online advertisements, mass emails, and in-person interactions at schools in various districts, including New Territories, Kowloon, and Hong Kong Island. Interested participants can enroll by completing an online application form using Qualtrics or Google form).

During offline recruitment sessions, staff will approach secondary school students and their parents (if the participants are under 18 years old) to obtain consent and have them complete a baseline questionnaire for further contact and intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

1. being a Hong Kong resident aged between 12-18 years;
2. having consumed alcohol in the past 12-month;
3. Using WhatsApp in their cell phone.

Exclusion Criteria:

1. cannot communicate in Cantonese or read Chinese;
2. currently using other alcohol control programs.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of drinking days | 3-month follow-up
  The primary outcome is the number of drinking days in the past 30 days at 3-month follow-up.

SECONDARY OUTCOMES:
Number of ever binge drinking days | 3-month follow-up
  Number of ever binge drinking days in the past 3 months at 3-month follow-up since trial participation
Number of binge drinking days | 3-month follow-up
  Number of binge drinking days in the past 30 days at 3-month
Intention to reduce or quit alcohol drinking | 3-month follow-up
  Intention to reduce or quit alcohol drinking in 10 points Likert scale at 3-month follow-up. [0: no intention | 10: Highest Intention]
Alcohol Use Disorder Identification Test | 3-month follow-up
  Alcohol Use Disorder Identification Test (AUDIT) score is a validated scale in measuring the impact of alcohol consumption on individual's health.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the completion of the relevant publications

REFERENCES:
- [Background] Garnett CV, Crane D, Brown J, Kaner EFS, Beyer FR, Muirhead CR, Hickman M, Beard E, Redmore J, de Vocht F, Michie S. Behavior Change Techniques Used in Digital Behavior Change Interventions to Reduce Excessive Alcohol Consumption: A Meta-regression. Ann Behav Med. 2018 May 18;52(6):530-543. doi: 10.1093/abm/kax029. PMID 29788261
- [Background] Wang H, Hu R, Zhong J, Du H, Fiona B, Wang M, Yu M. Binge drinking and associated factors among school students: a cross-sectional study in Zhejiang Province, China. BMJ Open. 2018 Apr 12;8(4):e021077. doi: 10.1136/bmjopen-2017-021077. PMID 29654047
- [Background] Ho DSY, Huang R, Wang MP, Lo WS, Lam TH. Adolescent alcohol drinking in Hong Kong: a school-based survey. Hong Kong Med J. 2019 Feb;25 Suppl 3(1):13-15. No abstract available. PMID 30792366
- [Background] Silveri MM. Adolescent brain development and underage drinking in the United States: identifying risks of alcohol use in college populations. Harv Rev Psychiatry. 2012 Jul-Aug;20(4):189-200. doi: 10.3109/10673229.2012.714642. PMID 22894728
- [Background] Hunt WA. Are binge drinkers more at risk of developing brain damage? Alcohol. 1993 Nov-Dec;10(6):559-61. doi: 10.1016/0741-8329(93)90083-z. PMID 8123218
- [Background] Zeigler DW, Wang CC, Yoast RA, Dickinson BD, McCaffree MA, Robinowitz CB, Sterling ML; Council on Scientific Affairs, American Medical Association. The neurocognitive effects of alcohol on adolescents and college students. Prev Med. 2005 Jan;40(1):23-32. doi: 10.1016/j.ypmed.2004.04.044. PMID 15530577
- [Background] Paljarvi T, Koskenvuo M, Poikolainen K, Kauhanen J, Sillanmaki L, Makela P. Binge drinking and depressive symptoms: a 5-year population-based cohort study. Addiction. 2009 Jul;104(7):1168-78. doi: 10.1111/j.1360-0443.2009.02577.x. Epub 2009 May 11. PMID 19438420
- [Background] Dahl RE. Adolescent brain development: a period of vulnerabilities and opportunities. Keynote address. Ann N Y Acad Sci. 2004 Jun;1021:1-22. doi: 10.1196/annals.1308.001. PMID 15251869
- [Background] Knight JR, Sherritt L, Harris SK, Gates EC, Chang G. Validity of brief alcohol screening tests among adolescents: a comparison of the AUDIT, POSIT, CAGE, and CRAFFT. Alcohol Clin Exp Res. 2003 Jan;27(1):67-73. doi: 10.1097/01.ALC.0000046598.59317.3A. PMID 12544008